CLINICAL TRIAL: NCT03416790
Title: IMPAACT 2015 - Evaluation of the HIV-1 Reservoir in the Central Nervous System of Perinatally-Infected Youth and Young Adults With Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IMPAACT 2015; DAIDS ID 35123 (Other: DAIDS CRMS)
Record Dates: First submitted 2018-01-18; First posted 2018-01-31 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: HIV-1-infection
Keywords: Central Nervous System; HIV Persistence; HIV Reservoirs

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — CSF, PBMC, plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
IMPAACT 2015 is a cross-sectional, exploratory study that will investigate the central nervous system (CNS) reservoir in perinatally HIV-infected adolescents and young adults on effective antiretroviral therapy with neurocognitive impairment. The study will assess the frequency with which HIV is detected in the cerebral spinal fluid (CSF) in this population and assess whether detectable HIV in the CSF correlates with markers of inflammation and neuronal injury. Findings from this study will advance understanding of the role of the CNS in HIV-1 persistence and its implications for future HIV-1 remission research.

DETAILED DESCRIPTION:
IMPAACT 2015 is a cross-sectional, exploratory study aiming to investigate the central nervous system (CNS) reservoir in perinatally HIV-infected adolescents and young adults on effective antiretroviral therapy with neurocognitive impairment. The study will assess the frequency with which HIV is detected in the cerebral spinal fluid (CSF) in this population and assess whether detectable HIV in the CSF correlates with markers of inflammation and neuronal injury. CSF will be examined for persistence of HIV-1 RNA or DNA despite antiretroviral therapy (ART) and for evidence of intrathecal inflammation. Perinatally-infected youth and young adults are of particular interest because there are very limited CSF data available in this population and reasons to be concerned about the CNS reservoir. In addition, measures of HIV-1 RNA in the CSF and associated biomarkers have not previously been explored in this population. A better understanding of viral persistence in the CSF, as well as CSF biomarker profiles, will provide preliminary data to move the field forward in understanding the role of the CNS in HIV-1 persistence and will have implications for future HIV-1 remission research.

ELIGIBILITY:
Inclusion Criteria:

* 13-24 years of age (inclusive) at enrollment (i.e., on the day the participant is enrolled in the study)
* Spoken fluency in English or Spanish
* If not of legal age to provide independent informed consent: Parent or legal guardian, or other legally authorized representative is willing and able to provide written informed consent for study participation and potential participant is willing and able to provide written assent for study participation
* If of legal age but not able to provide independent informed consent due to cognitive impairment as determined by site standard operating procedures (SOPs) and consistent with site institutional review board/ethics committee (IRB/EC) policies and procedures: Parent, legal guardian, or other legally authorized representative is willing and able to provide written informed consent for study participation and potential participant is willing and able to provide written assent for study participation
* If of legal age and able to provide independent informed consent as determined by site SOPs and consistent with site IRB/EC policies and procedures: Willing and able to provide written informed consent for study participation
* Has confirmed perinatal HIV-1 infection - with no documented evidence to suggest another route of transmission - based on review of available medical records
* Has been taking combination ART comprised of at least three agents from at least two classes of antiretroviral therapy for at least 12 consecutive months prior to enrollment as determined by the site investigator or designee based on participant or parent/guardian report and available medical records; regimen changes within the 12 months prior to enrollment are permitted, provided the virologic requirements in criterion below are met
* Has at least two consecutive documented plasma HIV-1 RNA values less than 40 copies/mL, at least three months apart, in the 12 months prior to enrollment; one of these values must be based on testing of a specimen collected within the 60 days prior to enrollment
* Has a Fluid Cognition Composite Score at least one-and-a-half standard deviations below the published normative mean (i.e., less than 78) based on administration of the NIH Toolbox Cognition Battery

Exclusion Criteria:

* Any ART interruption for more than seven consecutive days in the 12 months prior to enrollment
* Any HIV-1 RNA value greater than 200 copies/mL in the 12 months prior to enrollment
* Completed any of the NIH Toolbox subtests specified within 90 days prior to screening
* Any documented full scale intelligence quotient (IQ) score more than three standard deviations below the published normative mean (i.e., less than 55) or a Fluid Cognition Composite Score more than three standard deviations below the published normative mean (i.e., less than 55) based on administration of the NIH Toolbox Cognition Battery at screening
* Any documented diagnosis of autism spectrum disorder, schizophrenia, or other psychotic disorder
* Any known prior infection of the CNS that may be persistent or recurrent (e.g., cryptococcal meningitis, neurosyphilis)
* Any known non-HIV-related cause or significant contributing factor for cognitive impairment (e.g., birth injury, head injury, stroke, major or mild neurocognitive disorder due to a condition other than HIV) per Diagnostic and Statistical Manual of Mental Disorders 4th Edition (DSM-V) criteria
* Any known or suspected current contraindication to lumbar puncture
* Any current sensory or motor impairment severe enough to preclude participation in study evaluations (e.g., blindness, lack of upper limb control)
* If female and of reproductive potential (defined as having experienced menarche and having no documented history of a sterilization procedure), known or suspected pregnancy
* Any serious or otherwise clinically significant infection of the CNS or bloodstream (other than HIV-1 infection) within 30 days prior to enrollment
* Any live vaccine received within 30 days prior to enrollment
* Any other (non-live) vaccine received within 7 days prior to enrollment
* Received prolonged (more than 14 days) or high dose immunosuppressants within 30 days prior to enrollment (high dose would include >1 mg/kg prednisone (or equivalent) or any biologic immunosuppressant such as monoclonal antibody based therapy)
* Ever received any medication or other approved or investigational agent that may impact HIV-1 reservoirs, including but not limited to: HIV-1 vaccines, HIV-1 gene therapies, Anti-HIV-1 broadly neutralizing antibodies (e.g., VRC01), Anti-PD-1 or anti-PD-L1 antibody, Histone deacetylase inhibitors (e.g., vorinostat, romidepsin, panobinostat), Toll-like receptor agonists, Cytotoxic chemotherapies, Roxolitinib, and Sirolimus

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Perinatally HIV-1-infected youth and young adults (13-24 years of age) with cognitive impairment, on suppressive antiretroviral therapy, from study sites in the United States
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Prevalence of quantifiable cell-free HIV-1 RNA CSF | Within 30 Days of Screening Initiation
  Quantifiable cell-free HIV-1 RNA CSF defined as an HIV-1 RNA assay result of ≥20 copies/mL
Prevalence of detectable HIV-1 DNA in CSF cell pellets | Within 30 Days of Screening Initiation
  Detectable HIV-1 DNA in CSF cell pellets defined as an HIV-1 DNA assay result of ≥1 copy in the cell pellet obtained from ≥10 ml of CSF

SECONDARY OUTCOMES:
Concentrations of inflammatory and neuronal injury biomarkers in CSF | Within 30 Days of Screening Initiation
  Biomarkers to be evaluated include neopterin, neurofilament light chain (NFL), tyrosine (Y), lysine (K) and leucine (L) - 40kDa (YKL-40), interleukin (IL-6), C-reactive protein (CRP), interferon gamma-induced protein 10 (IP-10/CXCL10), monocyte chemoattractant protein 1 (MCP-1/CCL2), tumor necrosis factor (TNF-α), sCD14, soluble CD163 (sCD163), soluble intercellular adhesion molecule type 5 (sICAM-5) (immunoassays). Concentrations of each of these biomarkers in CSF will be summarized descriptively.
Concentrations of inflammatory and neuronal injury biomarkers in plasma | Within 30 Days of Screening Initiation
  Biomarkers to be evaluated include neopterin, neurofilament light chain (NFL), tyrosine (Y), lysine (K) and leucine (L) - 40kDa (YKL-40), interleukin (IL-6), C-reactive protein (CRP), interferon gamma-induced protein 10 (IP-10/CXCL10), monocyte chemoattractant protein 1 (MCP-1/CCL2), tumor necrosis factor (TNF-α), sCD14, soluble CD163 (sCD163), soluble intercellular adhesion molecule type 5 (sICAM-5) (immunoassays). Concentrations of each of these biomarkers in plasma will be summarized descriptively.
Associations of the above-listed secondary outcomes with the primary outcomes | Within 30 Days of Screening Initiation
  Associations will be assessed with Spearman correlations (and corresponding confidence intervals).

CONTACTS AND LOCATIONS:
Overall Officials: Ann Chahroudi, MD, PhD, Study Chair — Emory University; Thor Wagner, MD, Study Chair — University of Washington
Locations (12):
- United States (11):
  - University of Southern California (CRS 5048), Los Angeles, California
  - David Geffen School of Medicine at University of California, Los Angeles (CRS 5112), Los Angeles, California
  - University of California, San Diego Mother-Child-Adolescent HIV Program (CRS 4601), San Diego, California
  - University of Colorado, Denver (CRS 5052), Aurora, Colorado
  - Emory University School of Medicine (CRS 5030), Atlanta, Georgia
  - Johns Hopkins University (CRS 5092), Baltimore, Maryland
  - Boston Medical Center Pediatric HIV Program (CRS 5011), Boston, Massachusetts
  - Bronx-Lebanon Hospital Center (CRS 5114), The Bronx, New York
  - Jacobi Medical Center (CRS 5013), The Bronx, New York
  - St. Jude Children's Research Hospital (CRS 6501), Memphis, Tennessee
  - Seattle Children's Hospital (CRS 5017), Seattle, Washington
- University of Puerto Rico Pediatric HIV/AIDS Research Program (CRS 6601), San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No